CLINICAL TRIAL: NCT03931811
Title: Effects of Short Wave Diathermy Added on Dextrose Prolotherapy Injections in Osteoarthritis of the Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Hale Karapolat, Professor in Physical Medicine and Rehabilitation Department, Ege University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HDKnee
Record Dates: First submitted 2019-04-26; First posted 2019-04-30 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis; Prolotherapy; Hypertonic dextrose solution injections; Short-wave diathermy
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Prolotherapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short wave diathermy group (Experimental): Patients were randomized into 2 groups depending on their patient number, with odd numbers being recruited to SWD group, and even numbers to sham SWD group.
  Prolotherapy solutions were injected using 25 gauge needle, with solutions being 6 ml 25 % dextrose (3 ml 20% dextrose + 3 ml 30% dextrose) for intraarticular, and 20 ml 15% dextrose (10 ml 0,9% NaCl + 10 ml 30% dextrose) for periarticular.
  SWD group took short wave diathermy with specifications of 400 watt power output, 27.12 MHz frequency, 11.06m wave length, using condensators and electrodes of 12 cm diameter parallel to the knee for 20 minutes(Enraf-Nonius, Curapuls 970 Short wave diathermy device). Both groups took injections in the beginning of the therapy, 3rd week and 6th week, a total of 3 times. SWD or sham SWD therapy was given right after the injections, also for a total of 3 times.
  Interventions: Device: Short wave diathermy; Other: Prolotherapy
- Sham diathermy group (Sham Comparator): Patients were randomized into 2 groups depending on their patient number, with odd numbers being recruited to SWD group, and even numbers to sham SWD group.
  Prolotherapy solutions were injected using 25 gauge needle, with solutions being 6 ml 25 % dextrose (3 ml 20% dextrose + 3 ml 30% dextrose) for intraarticular, and 20 ml 15% dextrose (10 ml 0,9% NaCl + 10 ml 30% dextrose) for periarticular.
  Sham SWD group took 20 minutes of SWD therapy with device not working(Enraf-Nonius, Curapuls 970 Short wave diathermy device).
  Interventions: Other: Prolotherapy

INTERVENTIONS:
Device: Short wave diathermy — SWD group took short wave diathermy with specifications of 400 watt power output, 27.12 MHz frequency, 11.06m wave length, using condensators and electrodes of 12 cm diameter parallel to the knee for 20 minutes(Enraf-Nonius, Curapuls 970 Short wave diathermy device).
  Arms: Short wave diathermy group
Other: Prolotherapy — Prolotherapy solutions were injected to the knee by a blinded physician in the group, using 25 gauge needle, with solutions being 6 ml 25 % dextrose (3 ml 20% dextrose + 3 ml 30% dextrose) for intraarticular, and 20 ml 15% dextrose (10 ml 0,9% NaCl + 10 ml 30% dextrose) for periarticular. Injection points wwere defined as medial collateral ligaments, adhesion points of quadriceps tendon, adhesion points of patellar tendon, tuberositas tibia, pes anserinus, lateral collateral ligaments, coronal ligaments, medial and lateral tibia plateaus. Patients were blinded to their treatment groups
  Other Names: Hypertonic dextrose injections

SUMMARY:
Goal: To show the effects of short wave diathermy added on prolotherapy injections in osteoarthritis of the knee on pain, physical functioning and quality of life.

Material and Methods: 63 patients with osteoarthritis of the knee with Kellgren-Lawrence (K-L) class 2 or 3 were included in the study. Patients were randomized to two grous, first being dextrose prolotherapy+ short wave diathermy(SWD), and second being dextrose prolotherapy with sham SWD. Patients were injected with dextrose prolotherapy solutions in the beginning, 3rd and 6th week of the study, for a total of 3 times, and took 20 minutes of SWD after injection(true or sham). Western Ontorio and McMaster Universities Osteoarthritis Index (WOMAC), Visual Analogous Scale for pain(VAS) and Short Form Health Survey (SF-36)were applied before, after(6th week) and at the 3rd month of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were being between 45 and 75 years old, knee pain of 3 months or longer duration, and having OA of the knee compatible with Kellgren-Lawrance class 2 or 3

Exclusion Criteria:

* Patients using analgesics other than acetaminophen, having pregnancy, diabetes mellitus, infectious or inflammatory arthritis, hemophilia, knee prosthesis, history of knee injections in last 3 months or anticoagulant use, allergy to ingredients of the solutions, having cardiac pacemaker or other device, or metallic implants were exluded from the study.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2018-04-04 (Actual); Study Completion 2018-04-04 (Actual)

PRIMARY OUTCOMES:
Visual Analogous Scale(for the intensity of pain)(VAS) | 3 months
  VAS was used to assess the resting pain intensity of the subjects. Patients were asked to show their intensity of pain on a 10 cm long line, with 0 end being no pain, and 10 cm end being highest amount of pain possible. The distance between the mark and the 0 end was measured and the result was recorded as milimeters.

SECONDARY OUTCOMES:
Western Ontorio and McMaster Universities Osteoarthritis Index (WOMAC) | 3 months
  WOMAC is an index for the assessment of osteoarthritis consisting of 24 questions, with subscales being pain(5 questions), stiffness(2 questions) and physical functioning(17 questions). Turkish version of the test is expressed as a likert type scale, ranging from 0 to 4, with greater numbers expressing higher severity. The greater scores are associated with more severe disease
Short Form-36 (SF-36) | 3 months
  SF-36 is an index for the evaluation of quality of life in a broad range of patients. It consists of 8 domains: Physical function, bodily pain, role-physical, general health, vitality, social function, role-emotional, and mental health. Each domain is expressed separately, rather than a total score. All of the domains are given from 0 to 100 points, with greater values being associated with a better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege university school of medicine, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided